CLINICAL TRIAL: NCT04172142
Title: Comparison of Physical and Psychosocial Characteristics of Pectus Excavatum and Carinatum Patients With Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-17/15
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pectus Deformity; Physical Disability; Psychosocial Impairment
Keywords: Pectus Carinatum; Pectus Excavatum; Physical Impairment; Psychosocial Impairment
MeSH Terms: conditions — Pectus Carinatum; Funnel Chest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy individuals of similar age and sex who meet the inclusion criteria
- Pectus Excavatum: Individuals with pectus excavatum that meet the inclusion criteria
- Pectus Carinatum: Individuals with pectus excavatum that meet the inclusion criteria

SUMMARY:
Chest wall deformities are the development of ribs, cartilage and sternum that form the chest wall together with isolated or abnormalities of the musculoskeletal system. Pectus excavatum and carinatum deformities are most common. It is reported that individuals with this problem have posture and physical impairments, difficulty in psychosocial relations and decreased quality of life.Therefore, in this study, the investigators aimed to evaluated the physical and psychosocial characteristics of patients with pectus excavatum and carinatum compared with healthy controls.

DETAILED DESCRIPTION:
Pectus excavatum (PE) and pectus carinatum (PC) are the most common anterior chest-wall deformities. Both of these malformations predominantly affect males. They often coincide with the vulnerable life phase of puberty, a period characterized by great physical, social, and emotional changes. Outer appearance becomes a major issue for adolescents, and those who display a visible disfigurement may be put at a disadvantage, having to come to terms with a difference in their looks and having to face the risk of harassment by their peers. Patients with pectus deformities often experience feelings of shame and try to hide their chests. This can be reflected in the choice of clothing or poor body posture. Many patients even avoid social activities and sports. They are aware of the fact that their deformity is generally not considered attractive, and some regard it as an obstacle in future relationships. Reduced self-confidence and selfesteem appear to be rather common characteristics of PE patients. Recently, several authors have assessed the improvement of quality of life and body image following surgical repair of PE. Yet, little is known about the degree to which patients, differ from healthy individuals within the same age group. Steinmann et al observed reduced disease-specific and general health related quality in patients with a chest malformation. Body image was highly impaired in both PE and PC patients. However, the number of patients (71 PE, 19, PC, 82 healthy individuals) was not matched and was not evaluated physical function. Also, they evaluated patients with a high degree of preoperative deformity in this study. Therefore, the investigators aimed to evaluated the physical and psychosocial characteristics of patients with pectus excavatum and carinatum compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chest wall deformity by doctor
* Not having any chronic systemic and musculoskeletal diseases and injuries for healthy individuals

Exclusion Criteria:

* Having chronic systemic disease
* Genetic disease
* Being psychologically diagnosed
* Having additional musculoskeletal diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pectus Excavatum,Pectus Carinatum and Healthy Controls (10-18 years age)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
New York Posture Rating Chart | Baseline time
  The rating chart is used to assess 13 areas of the body, based on the assumption that posture is the alignment of the body and its segments. 13 regions (head, neck, shoulder, scapula, upper thoracic, waist, rips, abdomen, hips, knees, legs, feet and toes) are assessed in two different positions (lateral and posterior). A score is allocated to each area according to the position: 5 points to the correct position; 3 points for a slight deviation, and 1 point for a pronounced deviation. Total score is between 18-90 points. higher the points better the postural alignment
International Physical Activity Questionnaire-Short Form (IPAQ) in the assessment of physical activity. | Baseline time
  The questionnaire interrogates the last 7 days regarding the following activities: (1) Time (minutes) spent for vigorous physical activities (football, basketball, aerobics, or fast bicycling, heavy lifting, carrying loads, etc.), (2) Time (minutes) spent for moderate physical activities (carrying light load, bicycling at a regular pace, folk dances, bowling, tennis etc.), and (3) Time spent for walking and time spent for sitting in a day. Physical activity levels of the participants were classified into low [600 the metabolic equivalent of task (MET)-minute/week), moderate (600 to 3000 MET minute/week), and high (> 3000 MET- minute/week) activity groups based on total physical activity scores. higher the points better the physical activity.
Extended version of the Musculoskeletal Questionnaire (NMQ-E) | Baseline time
  The extended version of the musculoskeletal questionnaire is completed by self-administration or face to face interview and provides reliable information on the onset, prevalence and outcomes of musculoskeletal pain in nine body regions (the neck, shoulder, upper back, elbow, wrist/hand, low back, hip/ thigh, knee, ankle/foot). The NMQ-E interrogates ache, pain or discomfort experienced in the nine body parts to date, for the last 12 months, for the last four weeks and on the day of the administration,with binary choice questions (yes or no).The frequency of the answer yes is high and shows us that musculoskeletal pain is high and is a bad score.
Flexibility test | Baseline time
  bilateral sit-and-reach test: Sitting on the floor or a mat, legs straight and feet 8-12 inches apart, the person being tested reaches forward with the arms (hands overlapping). The distance of reach is measured in inches using a measuring line marked on the floor
Grip strength | Baseline time
  The test is conducted with the participant seated on a chair (with a back and no arm rests), with the lower limbs resting on the ground. The shoulder of the limb to be tested remained adducted and neutral for rotation, with the elbow flexed at 90 °, the forearm neutral and wrist extension between 0 and 30 ° with 0-15 degrees of ulnar deviation. During the test, constant verbal encouragement was given to the participants to use their maximum strength. The test is repeated three times to obtain the mean.
Abdominal muscle endurance | Baseline time
  Abdominal muscle endurance is measured as the number of correctly completed sit-ups in 30seconds. Sit-ups were performed with the hands placed at the side of the head, knees bent at 90°, and the feet secured by the investigator. A full sit-up is defined as touching the knees with the elbows and returning the shoulders to the ground. A higher number of completed sit-ups indicates greater abdominal muscle endurance.
Back strength | Baseline time
  Back strength of the participants is measured using a Back-leg-chest dynamometer. The participant was positioned with body erect and knees bent so that the grasping hand rests at proper height. Then, by straightening the knees and lifting the chain of the dynamometer, pulling force is applied on the handle. The body would be inclined forward at an angle of 60 degrees for the measurement of back strength
Social Appearance Anxiety Scale | Baseline time
  The scale a 16-item measure, was developed to assess the respondent's anxiety surrounding situations in which one's appearance may be evaluated. Response options for each item range from 1 (not at all) to 5 (extremely). The total score is calculated by summing across all items, after reverse coding the first item. Scores range from 16 to 80, with higher scores indicating greater fear
Pediatric Quality of Life Inventory (PedsQL), | Baseline time
  QoL was measured with one of the three age-appropriate versions (5-7, 8-12, 13-18 years). This scale measures children's perceptions and reflects their concerns on the dimensions of physical health (8 items) and psychosocial health, the latter comprising the subdimensions of emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). The overall QoL score is obtained by adding up the scores for all dimensions. Children were asked to indicate on a 3-point (5-7 year version) or 5-point (8 years and older versions) Likert scale to what extent they had experienced difficulties regarding these dimensions over the last month (0 = never, 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). The answers were reverse-scored and rescaled to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A score of 100 represents the best possible QoL, a score of 0 the worst.

SECONDARY OUTCOMES:
Brief Symptom Inventory | Baseline time
  This instrument measures the participant's subjective experience of symptoms during the last week and includes 53 items rated on five-point Likert scales ranging from 0 (not at all) to 4 (very much). Nine symptom dimensions (somatization, obsessive-compulsive behavior, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism) are assessed and reflected as subscales. The total score of the instrument represents the Global Severity Index used in this study as an indicator of patients' overall symptoms. Total brief symptom inventory score, and scores on subscales, are computed as the sum of item-scores divided by the number of items. Higher scores indicate more severe psychiatric symptoms.
Body Image Scale (BIS) | Baseline time
  Items of scale is associated a function ora part of the body. Each item has five possible choices as" I disagree strongly" , "I disagree" , "I am not sure", "I agree" and "I agree strongly". BIS item scores are from 1 to 5, total score varies between 40 and 200.A score of 135 and below from BIS is calculated as the body image is low

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, individual participant data will be shared with the authors every two months

REFERENCES:
- [Background] Akkas Y, Gulay Peri N, Kocer B, Gulbahar G, Baran Aksakal FN. The prevalence of chest wall deformity in Turkish children. Turk J Med Sci. 2018 Dec 12;48(6):1200-1206. doi: 10.3906/sag-1807-180. PMID 30541247
- [Background] Bahadir AT, Kuru P, Afacan C, Ermerak NO, Bostanci K, Yuksel M. Validity and reliability of the Turkish version of the nuss questionnaire modified for adults. Korean J Thorac Cardiovasc Surg. 2015 Apr;48(2):112-9. doi: 10.5090/kjtcs.2015.48.2.112. Epub 2015 Apr 5. PMID 25883894
- [Background] Banever GT, Konefal SH, Gettens K, Moriarty KP. Nonoperative correction of pectus carinatum with orthotic bracing. J Laparoendosc Adv Surg Tech A. 2006 Apr;16(2):164-7. doi: 10.1089/lap.2006.16.164. PMID 16646710
- [Background] Canavan PK, Cahalin L. Integrated physical therapy intervention for a person with pectus excavatum and bilateral shoulder pain: a single-case study. Arch Phys Med Rehabil. 2008 Nov;89(11):2195-204. doi: 10.1016/j.apmr.2008.04.014. PMID 18996250
- [Background] Blanco FC, Elliott ST, Sandler AD. Management of congenital chest wall deformities. Semin Plast Surg. 2011 Feb;25(1):107-16. doi: 10.1055/s-0031-1275177. PMID 22294949
- [Background] Hart TA, Flora DB, Palyo SA, Fresco DM, Holle C, Heimberg RG. Development and examination of the social appearance anxiety scale. Assessment. 2008 Mar;15(1):48-59. doi: 10.1177/1073191107306673. PMID 18258731
- [Background] Sahin NH, Durak Batigun A, Ugurtas S. [The validity, reliability and factor structure of the Brief Symptom Inventory (BSI)]. Turk Psikiyatri Derg. 2002 Summer;13(2):125-35. Turkish. PMID 12794665
- [Background] Einsiedel E, Clausner A. Funnel chest. Psychological and psychosomatic aspects in children, youngsters, and young adults. J Cardiovasc Surg (Torino). 1999 Oct;40(5):733-6. PMID 10597013
- [Background] Harkonen R, Piirtomaa M, Alaranta H. Grip strength and hand position of the dynamometer in 204 Finnish adults. J Hand Surg Br. 1993 Feb;18(1):129-32. doi: 10.1016/0266-7681(93)90212-x. PMID 8436850
- [Background] Lockie R, Schultz A, Callaghan S, Jordan C, Luczo T, Jeffriess M. A preliminary investigation into the relationship between functional movement screen scores and athletic physical performance in female team sport athletes. Biol Sport. 2015 Mar;32(1):41-51. doi: 10.5604/20831862.1127281. Epub 2014 Nov 3. PMID 25729149
- [Background] Kelly RE Jr, Cash TF, Shamberger RC, Mitchell KK, Mellins RB, Lawson ML, Oldham K, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Bagley T, Quinn A, Moskowitz AB. Surgical repair of pectus excavatum markedly improves body image and perceived ability for physical activity: multicenter study. Pediatrics. 2008 Dec;122(6):1218-22. doi: 10.1542/peds.2007-2723. PMID 19047237
- [Background] Roberts J, Hayashi A, Anderson JO, Martin JM, Maxwell LL. Quality of life of patients who have undergone the Nuss procedure for pectus excavatum: Preliminary findings. J Pediatr Surg. 2003 May;38(5):779-83. doi: 10.1016/jpsu.2003.50166. PMID 12720193
- [Background] Steinmann C, Krille S, Mueller A, Weber P, Reingruber B, Martin A. Pectus excavatum and pectus carinatum patients suffer from lower quality of life and impaired body image: a control group comparison of psychological characteristics prior to surgical correction. Eur J Cardiothorac Surg. 2011 Nov;40(5):1138-45. doi: 10.1016/j.ejcts.2011.02.019. Epub 2011 Mar 25. PMID 21440452
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] WELCH KJ. Satisfactory surgical correction of pectus excavatum deformity in childhood; a limited opportunity. J Thorac Surg. 1958 Nov;36(5):697-713. No abstract available. PMID 13588724